CLINICAL TRIAL: NCT01560299
Title: Evaluation of Optimal Time of Methimazole Discontinuation Before Radio-iodine Therapy in Hyperthyroid Grave's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, S.R.ZAKAVI, associate professor, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Metiodine
Record Dates: First submitted 2012-03-01; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Graves Disease
Keywords: hyperthyroidism; radio-iodine; I-131; methimazole; graves disease
MeSH Terms: conditions — Graves Disease; Hyperthyroidism | interventions — Methimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- group one (Active Comparator): This group will be advised to discontinue methimazole 24-48 hour before iodine therapy
  Interventions: Drug: Methimazole
- group two (Active Comparator): methimazole stopped 48-72 hour before radioiodine therapy
  Interventions: Drug: Methimazole
- group three (Active Comparator)
  Interventions: Drug: Methimazole

INTERVENTIONS:
Drug: Methimazole — Methimazole was stopped 24-48 before radio-iodine therapy
  Arms: group one
Drug: Methimazole — methimazole discontinued 49-72 hours before radioiodine treatment
  Arms: group two
Drug: Methimazole — methimazole discontinued 73-168 hours before radio-iodine treatment
  Arms: group three

SUMMARY:
Iodine therapy is the best treatment for graves disease.Most patients receive methimozale prior to radio-iodine treatment. This may decrease treatment response to iodine therapy.

Some physicians advice to discontinue methimazole 3 days before radioiodine therapy and others prefer longer off - methimazole period which bothers most patients. This study aimed to evaluate optimum time for methimazole discontinuation in graves disease.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* graves disease(TSH<0.1 &increased FT4 & positive TSI
* one or more bartlena criteria for radio-iodine therapy
* 24 hour RAIU>25%
* euthyroidism after methimazole treatment

Exclusion Criteria:

* pregnancy or lactation
* moderate or severe graves ophthalmopathy
* CHF or coronary heart disease
* palpable thyroid nodule
* lithium or amiodarone or lugol or ipodate treatment
* recent imaging with contrast agent
* very large goiter(more than 150 gram)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
thyroid function tests over one year after radioiodine therapy | months 1 , 3 ,6,9,12
  thyroid function test may change over one year . In order to consider the patients as cured ,thyroid function tests should reveal hypothyroidism or euthyroidism . In order to rule out temporary hypothyroidism the tests should be repeated after 6 months of radioiodine therapy.

CONTACTS AND LOCATIONS:
Overall Officials: rasoul zakavi, associate professor, Principal Investigator — Mashhad University of Medical Sciences
Locations (1):
- Mashad University of Medical Sciences, Mashhad, Khorasan Razavi, Iran